CLINICAL TRIAL: NCT02054897
Title: Efficacy and Safety of Semaglutide Once-weekly Versus Placebo in Drug-naïve Subjects With Type 2 Diabetes
Acronym: SUSTAIN™1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3623; 2013-000632-94 (EudraCT Number); U1111-1139-3090 (Other: WHO); JapicCTI-142442 (Registry Identifier: JAPIC)
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Semaglutide 1.0 mg (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide 0.5 mg (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide placebo 1.0 mg (Placebo Comparator)
  Interventions: Drug: placebo
- Semaglutide placebo 0.5 mg (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Once weekly, administrated subcutaneously (s.c. under the skin)
  Arms: Semaglutide 0.5 mg; Semaglutide 1.0 mg
Drug: placebo — Once weekly, administrated subcutaneously (s.c. under the skin)
  Arms: Semaglutide placebo 0.5 mg; Semaglutide placebo 1.0 mg

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate efficacy and safety of semaglutide once-weekly versus placebo in drug-naïve subjects with type 2 diabetes. (SUSTAIN™ 1-Monotherapy).

ELIGIBILITY:
Inclusion Criteria: - For Japan only: Male or female, age above or equal to 20 years at the time of signing inform consent - Subjects diagnosed with type 2 diabetes and treated with diet and exercise for at least 30 days before screening - HbA1c 7.0 - 10.0 % (53 - 86 mmol/mol) (both inclusive) Exclusion Criteria: - Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice) throughout the trial including the 5 week follow-up period. United Kingdom: Adequate contraceptive measures are defined as established use of oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device or intrauterine system, barrier methods of contraception (condom or occlusive cap with spermicidal foam/gel/film/cream/suppository), male sterilisation (where partner is sole partner of subject), or true abstinence (when in line with preferred and usual lifestyle) - Any chronic disorder or severe disease which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol - Treatment with any glucose lowering agent(s) in a period of 90 days prior to screening. An exception is short-term treatment (no longer than 7 days in total) with insulin in connection with inter-current illness - History of chronic or idiopathic acute pancreatitis - Screening calcitonin value above or equal to 50 ng/L (pg/mL) - Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 (MEN 2) - Impaired renal function defined as eGFR (estimated glomerular filtration rate ) below 30 mL/min/1.73 m^2 per modification of diet in renal disease (MDRD) formula (4 variable version) - Acute coronary or cerebrovascular event within 90 days before randomisation - Heart failure, New York Heart Association class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2015-05-08 (Actual); Study Completion 2015-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (76):
- United States (33):
  - Novo Nordisk Investigational Site, Anniston, Alabama
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Pell City, Alabama
  - Novo Nordisk Investigational Site, Hawaiian Gardens, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Miami Lakes, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Brownsburg, Indiana
  - Novo Nordisk Investigational Site, Franklin, Indiana
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Olive Branch, Mississippi
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Belvidere, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Delaware, Ohio
  - Novo Nordisk Investigational Site, Levittown, Pennsylvania
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Sealy, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
- Canada (7):
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Pointe-Claire, Quebec
  - Novo Nordisk Investigational Site, Trois-Rivières, Quebec
- Italy (6):
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Pisa
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Rome
  - Novo Nordisk Investigational Site, Siena
  - Novo Nordisk Investigational Site, Terni
- Japan (3):
  - Novo Nordisk Investigational Site, Kyoto-shi, Kyoto
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
- Mexico (3):
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
  - Novo Nordisk Investigational Site, Ciudad Madero, Tamaulipas
  - Novo Nordisk Investigational Site, Aguascalientes
- Romania (4):
  - Novo Nordisk Investigational Site, Oradea, Bihor County
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Buzău
  - Novo Nordisk Investigational Site, Galati
- Russia (8):
  - Novo Nordisk Investigational Site, Arkhangelsk
  - Novo Nordisk Investigational Site, Chelyabinsk
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saint-Petesburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Stavropol
- South Africa (8):
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Krugersdorp, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Vrededorp, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, eMkhomazi, KwaZulu-Natal
- United Kingdom (4):
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, St Helens
  - Novo Nordisk Investigational Site, Swansea

REFERENCES:
- [Background] Overgaard RV, Lindberg SO, Thielke D. Impact on HbA1c and body weight of switching from other GLP-1 receptor agonists to semaglutide: A model-based approach. Diabetes Obes Metab. 2019 Jan;21(1):43-51. doi: 10.1111/dom.13479. Epub 2018 Aug 23. PMID 30047216
- [Background] Fonseca VA, Capehorn MS, Garg SK, Jodar Gimeno E, Hansen OH, Holst AG, Nayak G, Seufert J. Reductions in Insulin Resistance are Mediated Primarily via Weight Loss in Subjects With Type 2 Diabetes on Semaglutide. J Clin Endocrinol Metab. 2019 Sep 1;104(9):4078-4086. doi: 10.1210/jc.2018-02685. PMID 30938762
- [Background] Rodbard HW, Bellary S, Hramiak I, Seino Y, Silver R, Damgaard LH, Nayak G, Zacho J, Aroda VR. GREATER COMBINED REDUCTIONS IN HbA1C >/=1.0% AND WEIGHT >/=5.0% WITH SEMAGLUTIDE VERSUS COMPARATORS IN TYPE 2 DIABETES. Endocr Pract. 2019 Jun;25(6):589-597. doi: 10.4158/EP-2018-0444. Epub 2019 Mar 13. PMID 30865526
- [Result] Sorli C, Harashima SI, Tsoukas GM, Unger J, Karsbol JD, Hansen T, Bain SC. Efficacy and safety of once-weekly semaglutide monotherapy versus placebo in patients with type 2 diabetes (SUSTAIN 1): a double-blind, randomised, placebo-controlled, parallel-group, multinational, multicentre phase 3a trial. Lancet Diabetes Endocrinol. 2017 Apr;5(4):251-260. doi: 10.1016/S2213-8587(17)30013-X. Epub 2017 Jan 17. PMID 28110911
- [Result] Warren M, Chaykin L, Trachtenbarg D, Nayak G, Wijayasinghe N, Cariou B. Semaglutide as a therapeutic option for elderly patients with type 2 diabetes: Pooled analysis of the SUSTAIN 1-5 trials. Diabetes Obes Metab. 2018 Sep;20(9):2291-2297. doi: 10.1111/dom.13331. Epub 2018 Jun 7. PMID 29687620
- [Result] Petri KCC, Ingwersen SH, Flint A, Zacho J, Overgaard RV. Exposure-response analysis for evaluation of semaglutide dose levels in type 2 diabetes. Diabetes Obes Metab. 2018 Sep;20(9):2238-2245. doi: 10.1111/dom.13358. Epub 2018 Jun 15. PMID 29748996
- [Result] Ahren B, Atkin SL, Charpentier G, Warren ML, Wilding JPH, Birch S, Holst AG, Leiter LA. Semaglutide induces weight loss in subjects with type 2 diabetes regardless of baseline BMI or gastrointestinal adverse events in the SUSTAIN 1 to 5 trials. Diabetes Obes Metab. 2018 Sep;20(9):2210-2219. doi: 10.1111/dom.13353. Epub 2018 Jun 12. PMID 29766634
- [Result] DeVries JH, Desouza C, Bellary S, Unger J, Hansen OKH, Zacho J, Woo V. Achieving glycaemic control without weight gain, hypoglycaemia, or gastrointestinal adverse events in type 2 diabetes in the SUSTAIN clinical trial programme. Diabetes Obes Metab. 2018 Oct;20(10):2426-2434. doi: 10.1111/dom.13396. Epub 2018 Jul 9. PMID 29862621
- [Result] Carlsson Petri KC, Ingwersen SH, Flint A, Zacho J, Overgaard RV. Semaglutide s.c. Once-Weekly in Type 2 Diabetes: A Population Pharmacokinetic Analysis. Diabetes Ther. 2018 Aug;9(4):1533-1547. doi: 10.1007/s13300-018-0458-5. Epub 2018 Jun 15. PMID 29907893
- [Result] Aroda VR, Ahmann A, Cariou B, Chow F, Davies MJ, Jodar E, Mehta R, Woo V, Lingvay I. Comparative efficacy, safety, and cardiovascular outcomes with once-weekly subcutaneous semaglutide in the treatment of type 2 diabetes: Insights from the SUSTAIN 1-7 trials. Diabetes Metab. 2019 Oct;45(5):409-418. doi: 10.1016/j.diabet.2018.12.001. Epub 2019 Jan 4. PMID 30615985
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- [Derived] DeSouza C, Cariou B, Garg S, Lausvig N, Navarria A, Fonseca V. Efficacy and Safety of Semaglutide for Type 2 Diabetes by Race and Ethnicity: A Post Hoc Analysis of the SUSTAIN Trials. J Clin Endocrinol Metab. 2020 Feb 1;105(2):dgz072. doi: 10.1210/clinem/dgz072. PMID 31769496
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 87 sites, selected for recruitment, 72 sites in 8 countries randomised subjects: Canada: 7 sites; Italy: 6 sites; Japan: 5 sites; Mexico: 2 sites; Russian Federation: 8 sites; South Africa: 8 sites; United Kingdom: 4 sites; United States: 32 sites.
Groups:
- Semaglutide 0.5 mg: Subjects were given 0.25 mg semaglutide once weekly subcutaneous (s.c.; under the skin) injections for 4 weeks followed by 0.5 mg semaglutide once weekly for the remaining 26 weeks of the treatment period.
- Semaglutide 1.0 mg: Subjects were given 0.25 mg semaglutide once weekly s.c. injection for 4 weeks, 0.5 mg semaglutide once weekly s.c. injections for the next 4 weeks followed by 1.0 mg semaglutide once weekly s.c. injections for the remaining 22 weeks of the treatment period.
- Placebo: Subjects were randomised to either of the 2 placebo arms (i.e., semaglutide placebo 0.5 mg and semaglutide placebo 1.0 mg) and then pooled for data analysis.
  1. Placebo 0.5 mg arm: Subjects were given 0.25 mg placebo once weekly s.c. injections for 4 weeks followed by 0.5 mg placebo once weekly s.c. injections for the remaining 26 weeks of the treatment period.
  2. Placebo 1.0 mg arm: Subjects were given 0.25 mg placebo once weekly s.c. injections for 4 weeks, 0.5 mg placebo once weekly s.c. injections for the next 4 weeks followed by 1.0 mg placebo once weekly s.c. injections for the remaining 22 weeks of the treatment period.
Period: Overall Study
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Started | 129 | 130 | 129
Exposed | 128 | 130 | 129
Completed | 119 | 123 | 117
Not Completed | 10 | 7 | 12
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Missing follow-up information | 3 | 5 | 3
Not completed — Lost to Follow-up | 4 | 2 | 7
Not completed — Randomized but not exposed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised subjects who had received at least 1 dose of randomised semaglutide (s.c.) or placebo.
Groups:
- Semaglutide 0.5 mg: Subjects were given 0.25 mg semaglutide once weekly s.c. injection for 4 weeks followed by 0.5 mg semaglutide once weekly s.c. injections for the remaining 26 weeks of the treatment period.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo | Total
Number analyzed (Participants) | 128 | 130 | 129 | 387
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (11.1) | 52.7 (11.9) | 53.9 (11.0) | 53.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 50 | 59 | 177
  Male | 60 | 80 | 70 | 210
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.09 (0.89) | 8.12 (0.81) | 7.95 (0.85) | 8.05 (0.85)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] — Population: Number of subjects analysed=subjects with data available for fasting plasma glucose at baseline.
  mmol/L
    number analyzed (Participants) | 125 | 129 | 127 | 381
    (all) | 9.66 (2.77) | 9.90 (2.50) | 9.68 (2.77) | 9.75 (2.67)
Body weight [Mean (Standard Deviation); unit: kilogram(s)] | 89.81 (22.96) | 96.87 (25.59) | 89.05 (22.16) | 91.93 (23.83)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 79.52 (9.06) | 79.25 (8.52) | 79.14 (8.39) | 79.30 (8.64)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 127.87 (13.15) | 128.89 (12.92) | 129.57 (13.50) | 128.78 (13.18)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline (week 0) in HbA1c was evaluated after 30 weeks of treatment. Missing data were imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: Week 0, week 30
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 128 | 130 | 129
Percentage of HbA1c | -1.47 (1.02) | -1.56 (1.26) | -0.00 (0.90)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Placebo; For the primary HbA1c endpoint, superiority was planned to be tested for semaglutide 1.0 mg versus placebo. The post-baseline responses were analysed using a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority — Superiority for change in HbA1c was claimed if the upper limit of the 2-sided 95% confidence interval (CI) for the estimated difference was below 0%; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.53, 95% CI 2-sided [-1.81 to -1.25] — Semaglutide 1.0 mg minus Placebo
Statistical Analysis 2: Comparison: Semaglutide 0.5 mg vs Placebo; For the primary HbA1c endpoint, superiority was planned to be tested for semaglutide 0.5 mg versus placebo, if superiority for semaglutide 1.0 mg was concluded. The post-baseline responses were analysed using a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority — Superiority for change in HbA1c was claimed if the upper limit of the 2-sided 95% CI for the estimated difference was below 0%; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.43, 95% CI 2-sided [-1.71 to -1.15] — Semaglutide 0.5 mg minus Placebo

2. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) in body weight was evaluated after 30 weeks of treatment. Missing data were imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: Week 0, week 30
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: kilogram(s)
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 128 | 130 | 129
kilogram(s) | -3.68 (4.03) | -4.67 (5.19) | -0.89 (3.46)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG was evaluated after 30 weeks of treatment. Missing data were imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: Week 0, week 30
Population: Full analysis set. Number of subject analysed=subjects who contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 125 | 129 | 127
mmol/L | -2.41 (2.55) | -2.39 (2.74) | -0.55 (2.2)

4. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: Change from baseline (week 0) in systolic and diastolic blood pressure was evaluated after 30 weeks of treatment. Missing data were imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: Week 0, week 30
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 128 | 130 | 129
mmHg
  Systolic blood pressure | -2.29 (12.58) | -2.74 (11.58) | -2.01 (11.23)
  Diastolic blood pressure | -0.73 (6.88) | 0.22 (7.6) | 0.60 (7.59)

5. Secondary Outcome: Subjects Who Achieve (Yes/no):HbA1c Below 7.0% (53 mmol/Mol) American Diabetes Association Target
Description: Percentage of subjects who achieve (yes/no): HbA1c below 7.0% (53 mmol/mol) American Diabetes Association target after 30 weeks' treatment. Missing HbA1c data imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: At 30 weeks of treatment
Population: Full analysis set
Measure: Number; unit: Percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 128 | 130 | 129
Percentage of subjects
  Yes | 74.2 | 72.3 | 24.8
  No | 25.8 | 27.7 | 75.2

6. Secondary Outcome: Subjects Who Achieve (Yes/no):HbA1c Below or Equal to 6.5% (48 mmol/Mol) American Association of Clinical Endocrinologists Target
Description: Percentage of subjects who achieve (yes/no): HbA1c below 6.5% (48 mmol/mol) American Diabetes Association target after 30 weeks' treatment. Missing HbA1c data imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: At 30 weeks of treatment
Population: Full analysis set
Measure: Number; unit: Percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 128 | 130 | 129
Percentage of subjects
  Yes | 59.4 | 60.0 | 13.2
  No | 40.6 | 40.0 | 86.8

ADVERSE EVENTS:
Time Frame: From the first trial product administration (in week 0) till the date of the end-of-treatment follow-up visit (in week 35 + the 7-day visit window) or on the date of the last trial product administration plus 42 days (5 weeks plus the 7 days visit window)
Description: Safety analysis set (SAS) included all randomised subjects who had received at least 1 dose of randomised semaglutide or placebo.
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 7/128 | 7/130 | 5/129
Other Adverse Events (participants affected / at risk) | 53/128 | 47/130 | 27/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=128) | Semaglutide 1.0 mg (N=130) | Placebo (N=129)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=128) | Semaglutide 1.0 mg (N=130) | Placebo (N=129)
Constipation (Gastrointestinal disorders) | 8 (9) | 5 (5) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 16 (27) | 14 (19) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 7 (13) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 15 (43) | 9 (18) | 8 (13)
Lipase increased (Investigations) | 8 (10) | 5 (5) | 5 (5)
Nasopharyngitis (Infections and infestations) | 6 (7) | 6 (9) | 7 (9)
Nausea (Gastrointestinal disorders) | 26 (44) | 31 (46) | 10 (12)
Vomiting (Gastrointestinal disorders) | 5 (11) | 9 (15) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property